CLINICAL TRIAL: NCT01230723
Title: RANDOMIZED TRIAL OF ZOTAROLIMUS- AND EVEROLIMUS-ELUTING STENTS REGARDING STENT COVERAGE ASSESSED BY OCT
Brief Title: Test Safety and Efficacy of Zotarolimus- and Everolimus-Eluting Stents (ZES/EES) Assessed by Optical Coherence Tomography
Acronym: ZES/EES-OCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S03210
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Everolimus-Eluting Stent
  Interventions: Device: Everolimus-Eluting-Stent
- Arm 2 (Active Comparator): Zotarolimus-Eluting-Stent
  Interventions: Device: Zotarolimus-Eluting-Stent

INTERVENTIONS:
Device: Everolimus-Eluting-Stent — due randomization everolimus-eluting-stent will be implanted
  Other Names: Xience-V®
  Arms: Arm 1
Device: Zotarolimus-Eluting-Stent — due randomization zotarolimus-eluting-stent will be implanted
  Other Names: Endeavor Resolute®
  Arms: Arm 2

SUMMARY:
The objective of the study is to assess the superiority of the everolimus-eluting stent (Endeavor Resolute®) compared with the everolimus-eluting stent (XIENCE V®) regarding uncovered stent strut segments.

DETAILED DESCRIPTION:
The mid-term efficacy of drug-eluting stents has been well-established, but there is an ongoing debate on the potential of an increased incidence of late stent thrombosis, particularly after discontinuation of thienopyridine therapy, as well as of delayed onset of restenosis or catch-up phenomenon with permanent polymer-based DES. The extent of strut coverage with reduction of exposed thrombogenic material has been shown to be associated with the inflammatory reaction grade and with the incidence of stent thrombosis. The optical coherence tomography (OCT) is an intravascular imaging modality based on light. The principle is similar to intravascular ultrasound, but due to the much shorter wave length of light, it offers a much better resolution up to 10µm, enabling the exact determination of strut coverage, neointimal thickness, vessel size, presence of dissections, and even the presence of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% stenosis located in native coronary vessels.
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
* In women with childbearing potential a negative pregnancy test is mandatory.

Exclusion Criteria:

* Lesion length >16mm requiring a stent length >18mm
* Target lesion located in the left main trunk.
* In-stent restenosis.
* Acute myocardial infarction
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Known allergy to the study medications: everolimus, zotarolimus, stainless steel or cobalt chrome.
* Inability to take dual antiplatelet therapy for at least 6 months.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Degree of stent strut coverage assessed by OCT for each visible strut segment | 6-8 months

SECONDARY OUTCOMES:
Percentage of malapposed strut assessed by OCT | 6-8 months
Percentage of uncovered malapposed struts assessed by OCT | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Tiroch, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - Klinikum rechts der Isar, Munich, Bavaria